CLINICAL TRIAL: NCT02770469
Title: Behavioral Intervention to Reduce Breast Cancer Disparity Among Underserved Koreans
Brief Title: Culturally Tailored Educational and Support Program to Increase Quality of Life Among Korean Breast Cancer Survivors
Acronym: TOGETHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R21CA178471 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Korean Americans; Survivorship; Quality of Life; Coping Skills; Perceived Stress
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Standard Intervention (Active Comparator): The standard intervention group received linguistically and culturally tailored information regarding breast cancer and survivorship.
  Interventions: Behavioral: Linguistically and Culturally Tailored Information
- Enhanced Intervention (Experimental): The enhanced intervention group received linguistically and culturally tailored information regarding breast cancer and survivorship as well as cognitive-behavioral stress management.
  Interventions: Behavioral: Linguistically and Culturally Tailored Information; Behavioral: Cognitive-Behavioral Stress Management

INTERVENTIONS:
Behavioral: Linguistically and Culturally Tailored Information — Participants received linguistically and culturally tailored information on diet and nutrition, physical activity, managing treatment side effects, follow-up care plans, complementary and alternative medicine, reducing environmental exposure to estrogen, navigating cancer-related financial issues, family history, body image, sexuality, and advances in breast cancer research.
Behavioral: Cognitive-Behavioral Stress Management — Participants learned and practiced skills related to mindfulness, relaxation, stress reduction, rational thinking, improving coping, enhancing social support, anger management, and assertiveness training.
  Arms: Enhanced Intervention

SUMMARY:
The objective of the TOGETHER (Together Overcome and Get Empowered Through Health Education and Relationships) program was to examine the effectiveness of one of the first linguistically and culturally tailored intervention programs to increase quality of life among Korean American breast cancer survivors.

DETAILED DESCRIPTION:
This study employed a randomized trial design, consisting of a standard and enhanced intervention group. Participants attended seven weekly sessions and one follow-up session that lasted for about 2 hours each. All sessions were conducted by two Korean female bilingual licensed clinical psychologists.

The specific aims of this study were to: (1) Implement and evaluate the effects of tailored intervention on perceived stress, coping and quality of life among Korean American breast cancer survivors; and (2) Conduct a process evaluation to assess the feasibility and fidelity of the intervention, which will provide data that can inform the development of future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Living in Maryland, Northern Virginia, or the Washington D.C. metropolitan area
* Have been diagnosed with breast cancer
* Have had surgery, completed treatment within the last two years, or still receiving adjuvant therapies

Exclusion Criteria:

* Unable to understand Korean

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Breast (FACT-B) | changes in quality of life during baseline, 7 weeks, and 14 weeks

SECONDARY OUTCOMES:
Cancer Behavior Inventory- Brief Version (CBI-B) | changes in self-efficacy for coping with cancer during baseline, 7 weeks, and 14 weeks
Perceived Stress Scale (PSS) | changes in stress during baseline, 7 weeks, and 14 weeks
Additional items to assess improvement in skills/knowledge covered by the intervention program | changes in responses during baseline, 7 weeks, and 14 weeks
  Participants were asked 12 multiple choice items on coping with stress, utilizing social support, anger management, assertiveness, and communicating with healthcare providers as well as 1 open-ended item on how participants cope with stress. Multiple choice items were on a 5-point Likert scale ranging from never to very often.

CONTACTS AND LOCATIONS:
Overall Officials: Sunmin Lee, ScD, Principal Investigator — University of Maryland School of Public Health

REFERENCES:
- See also: TOGETHER Program website — https://www.togetherprogram.org/